CLINICAL TRIAL: NCT03469869
Title: The Effect of Balanced and Sustainable Diet for Insulin Resistance and Inflammation Marker of Obese Adults in Indonesia
Brief Title: Effects of Balanced and Sustainable Diet Application for Insulin Resistance and Inflammation Marker of Obese People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Rina Agustina, Head of Human Nutrition Research Center, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YULIA-SAMI project
Record Dates: First submitted 2018-02-27; First posted 2018-03-19 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Insulin Resistance; Inflammation; Blood Glucose, High
Keywords: Obesity
MeSH Terms: conditions — Obesity; Insulin Resistance; Inflammation

STUDY DESIGN:
Intervention Model Description: One group balance diet One group balance and sustainable diet
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Giving a spesific personal menu through android apps, one group with balance diet menu, and the other with balance and sustainable diet menu. Only di IT knows which person get which type of menu
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- balanced and sustainable diet (Experimental): The intervention group will receive menu recommendation of restriction calorie balanced and sustainable diet for 8 weeks. the control group will receive menu recommendation of balanced diet for 8 weeks. these menus are given in the apps
  Interventions: Other: balanced and sustainable diet
- balanced diet (Active Comparator): the intervention group receive get menu recommendation of restriction calorie balanced and sustainable diet for 8 weeks. the other group will receive menu recommendation of balanced diet for 8 weeks. these menus are given in the apps
  Interventions: Other: balanced and sustainable diet

INTERVENTIONS:
Other: balanced and sustainable diet — the intervention group will get menu recommendation of restriction calorie balanced and sustainable diet for 8weeks. the other group will get menu recommendation of balanced diet for 8 weeks. these menus are given in the apps named EatsUp.
  the intervention group will get menu recommendation of restriction calorie balanced and sustainable diet for 8 weeks. the other group will get menu recommendation of balanced diet for 8 weeks. these menus are given in the apps named EatsUp.

SUMMARY:
This study evaluates the effect of balanced and sustainable diet application on fat composition, insulin resistance and inflammation marker in obese people.

Intervention: Obese subject will receive intervention on balanced and sustainable diet application Control: Obese subject will receive a balanced diet application only

DETAILED DESCRIPTION:
Maintaining the adherence of weight loss programme while selecting healthy and sustainable foods will become a worldwide future challenge in nutrition. Therefore, we investigated the suitable content, graphic, and flow in developing a mobile application as an alternative solution for enhancing the compliance of weight control and selecting healthy food with the least environmental impact.

The treatment for obesity consists of dieting, physical exercise, pharmacology, and surgery. Restricted balanced diet is a well known diet recommendation for people with obesity. Sustainable diet is an alternative form of diet which contributes to healthy life and is protective of biodiversity.

The main challenge in obesity management is the sustainability of weight loss programme. Mobile apps are an alternative solution for enhancing compliance.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 25 kg/m2
* using Android-based smartphone
* willing to join this research by signing informed consent

Exclusion Criteria:

* pale in physical examination
* in weight loss program
* have obesity with comorbidities
* have hormonal diseases
* consumed hormonal drug, PTU, anti diabetes drug
* smoking or stop smoking under 2 years
* pregnant and breastfeeding women

Ages: 19 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Change of body weight | baseline at Day0 and endline at Day56
  Change from baseline body weight at 8 weeks, is measured in kg

SECONDARY OUTCOMES:
Change of Fat Mass | baseline at Day0 and endline at Day56
  Change from baseline Fat Mass at 8 weeks, is measured by body composition analyzer in kg
Change of Fasting plasma glucose | baseline at Day0 and endline at Day56
  Change from baseline Fasting plasma glucose at 8 weeks, is measured in mg/dL
Change of TNF alpha | baseline at Day0 and endline at Day56
  Change from baseline TNF alpha at 8 weeks, is measured in pg/ml
Change of Fasting Insulin | baseline at Day0 and endline at Day56
  Change from baseline Fasting Insulin at 8 weeks, is measured in µU/mL
Change of HOMA-IR | baseline at Day0 and endline at Day56
  Change from baseline HOMA-IR at 8 weeks, is measured using formulation : glukosa (mg/dL) x insulin (µU/mL)/405
Change of Waist Circumference | baseline at Day0 and endline at Day56
  Change from baseline Waist Circumference at 8 weeks, is measured in cm
Change of Carbohydrate intake | baseline at Day0 and endline at Day56
  Change from baseline Carbohydrate intake at 8 weeks, is measured in gram using 24HR-recall
Change of Fat intake | baseline at Day0 and endline at Day56
  Change from baseline Fat intake at 8 weeks, is measured in gram using 24HR-recall
Change of Protein intake | baseline at Day0 and endline at Day56
  Change from baseline Protein intake at 8 weeks, is measured in gram using 24HR-recall

CONTACTS AND LOCATIONS:
Overall Officials: Rina Agustina, PhD, Principal Investigator — Indonesia University
Locations (1):
- University of Indonesia, Depok, West Java, Indonesia

REFERENCES:
- [Derived] Agustina R, Febriyanti E, Putri M, Martineta M, Hardiany NS, Mustikawati DE, Hanifa H, Shankar AH. Development and preliminary validity of an Indonesian mobile application for a balanced and sustainable diet for obesity management. BMC Public Health. 2022 Jun 20;22(1):1221. doi: 10.1186/s12889-022-13579-x. PMID 35725407